CLINICAL TRIAL: NCT02837588
Title: Endocavitary Radiofrequency Treatment in Patients Who Present With Chronic Pelvic Pain Compared to Usual Drug Therapy
Brief Title: Hyperthermy Endocavitary Treatment in Pelvic Pain
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Hospital Universitario Virgen de la Victoria (Other)
Responsible Party: Principal Investigator, Marta Jerez Sainz, Director, coordinator of Pelvic floor department, Principal Investigator, Clinical Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyperthermy pelvic floor
Record Dates: First submitted 2016-07-06; First posted 2016-07-19 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Pelvic Pain
Keywords: chronic pelvic pain; trigger points; hiperthermy
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperthermy treatment with MJS electrode (Active Comparator): 30 patients who are diagnosed with myofascial syndrome by gyneacologist or urologist goes to Pelvic Floor Physiotherapist for 4 session with hyperthermy treatment with MJS electrode at pelvic floor trigger points
  Interventions: Device: Hyperthermy treatment with MJS electrode
- CONTROL (No Intervention): No intervention with radiofrequency treatment, only evaluation to usual drug treatment

INTERVENTIONS:
Device: Hyperthermy treatment with MJS electrode — 30 patients who are diagnosed Pelvic pain with myofascial syndrome by gyneacologist or urologist goes to Pelvic Floor Physiotherapist for 4 session with hyperthermy treatment with MJS electrode at pelvic floor trigger points
  Arms: Hyperthermy treatment with MJS electrode

SUMMARY:
* Treatment at pelvic floor with hyperactivity with hyperthermy electrode MJS
* MJS electrode is effective for transvaginal treatment at pelvic pain patients
* Hyperthermy treatment with MJS electrode is more effective to usual drugs treatment

DETAILED DESCRIPTION:
This study analyzed the evolution of chronic pelvic pain, defined by the different map of myofascial trigger points assets presents the patient with medical treatment compared to treatment with radiofrequency endocavitary electrode MJS. The initial evaluator analyzed by the NIH-CPSI Scale questionnaire and symptoms of chronic pelvic pain Stanford Protocol for female or male quality of life of the patient before the doctor or radio frequency and a month since treatment. the patient to the Principal Investigator, specialist physiotherapist, who appreciates tenderness the presence of a taut band with a map of pain in endopelvic and exopelvic muscles, determining the activation of myofascial trigger points in each is derived. The Principal Investigator proceeds to address each active myofascial trigger points with the MJS electrode four 20-minute sessions twice a week. The MJS has a curved end pressure which favors the compression point plus the location and accurate approach Radiofrequency pathological point as outstanding feature. The high specificity of myofascial treatment offered by the MJS electrode involves no danger, besides having the computer screen conductivity meter and a temperature sensor on the head to control both parameters in real time during the treatment session

ELIGIBILITY:
Inclusion Criteria:

* Women with chronic pelvic pain

Exclusion Criteria:

* chronic pelvic pain or neurological degenerative etiology
* Presence of pathology or infectious processes genitourinary level
* possibility of pregnancy or lactating.
* Lack of informed consent, mental disorders, dementia, dependent people who need tutor.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
NIH-CPSI questionnaire | four weeks
  questions for pelvic pain evaluation

SECONDARY OUTCOMES:
pain measure questionnaire | four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Walker, Dr, Study Director — Universitat Central de Catalunya; Marta Losa, Dr, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Marta Sainz, Málaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes
It's approved from 2015 May to 2016 December, when the investigators have to report clinical trial conclusions